CLINICAL TRIAL: NCT07029659
Title: A Study Evaluating the Diagnostic Performance of OCS in the Differential Diagnosis of Endometriosis vs. Endometriosis-Associated Ovarian Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PekingUMCH-OCS
Record Dates: First submitted 2025-06-11; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-01

CONDITIONS: Endometriosis; Endometriosis-Associated Ovarian Carcinoma
Keywords: Endometriosis; EAOC; OCS score
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ovarian Cancer Score — Preoperatively, 5 ml blood samples were collected for OCS testing to determine the benign or malignant nature of ovarian endometriotic tissues. The OCS results were statistically analyzed against the gold standard of histopathological diagnosis.

SUMMARY:
Prospectively enroll patients with endometriosis and EAOC who complete the routine diagnostic and treatment process and consent to surgical intervention for OCS testing. Using postoperative ovarian pathological diagnosis as the gold standard, evaluate the clinical diagnostic performance of exosome detection in differentiating between endometriosis and EAOC.

ELIGIBILITY:
Inclusion Criteria:

* (1) Females aged ≥18 years; (2) Initial diagnosis of endometriosis or EAOC based on clinical presentation and imaging findings (including transvaginal ultrasound and MRI), with surgical indications; (3) Consent to surgical treatment and availability of postoperative ovarian pathological diagnosis; (4) Sufficient specimens for serum marker testing; (5) Voluntary participation in this study with signed informed consent form.

Exclusion Criteria:

* (1) Pregnant and lactating women; (2) Patients who have previously undergone surgery with available ovarian histopathological examination results; (3) Confirmed cases of recurrent ovarian carcinoma; (4) Patients receiving chemotherapy or pelvic radiotherapy within 6 months prior to sample collection; (5) Concurrent primary malignancies; (6) Contraindications to surgical evaluation or inability to obtain ovarian surgical pathology information; (7) Specimens non-conforming to collection/preservation requirements, or contaminated/suspected contaminated samples.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Endometriosis and Endometriosis-Associated Ovarian Carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 336 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The diagnostic performance of OCS in distinguishing EAOC from benign endometriotic lesions, including sensitivity and specificity. | Preoperative blood draw.

SECONDARY OUTCOMES:
The diagnostic performance of OCS for early-stage EAOC; its performance in differentiating various types of endometriosis and distinguishing EAOC subtypes. | Preoperative blood draw.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital (PuMCH), Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Sharing research findings through article publication
Supporting Information: Study Protocol, ICF